CLINICAL TRIAL: NCT03293329
Title: Effects of Diaphragm Muscle Therapy on Pain and Shoulder Movement in Subjects With Rotator Cuff Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Isidro Fernández López, Principal Investigator, Universidad Complutense de Madrid
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: UComplutenseMadrid Fasisifer1; 2017-003316-39 (EudraCT Number)
Record Dates: First submitted 2017-09-16; First posted 2017-09-26 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Rotator Cuff Injury; Diaphragm; Relaxation
Keywords: rotator cuff injury; diaphragm; physical therapy; manual therapy
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diaphragm manual therapy (Experimental): 3 diaphragm stretching techniques performed by a physical therapist are employed in this experimental group during 10 minutes. The participants are situated in a seated, supine and side bending position. 20 people are recruited in order to the inclusion criteria for the study. They have rotator cuff injuries diagnosed by ultrasounds or magnetic resonance.
  Interventions: Other: Diaphragm manual therapy techniques
- Diaphragm hipopressive exercise (Experimental): Diaphragm mobilization through active hipopressive gymnastic exercise in two different postures. 20 people are recruited in order to the inclusion criteria for the study. They have rotator cuff injuries diagnosed by ultrasounds or magnetic resonance.
  Interventions: Other: Diaphragm mobilization through active hipopressive gymnastic exercise
- Shoulder myofascial trigger points treatment (Active Comparator): A ischemic compression technique in infraespinatus and supraespinatus myofascial trigger points performed by a physical therapist is employed in this group. 20 people are recruited in order to the inclusion criteria for the study. They had rotator cuff injuries diagnosed by ultrasounds or magnetic resonance.
  Interventions: Other: Ischemic compression techniques in shoulder myofascial trigger points

INTERVENTIONS:
Other: Diaphragm manual therapy techniques — 3 diaphragm manual therapy techniques performed by a physical therapist are employed in this experimental group during 10 minutes. The participants are situated in a seated, supine and side bending position.
  Arms: Diaphragm manual therapy
Other: Diaphragm mobilization through active hipopressive gymnastic exercise — Diaphragm mobilization through active hipopressive gymnastic exercise in two different postures: standing and standing bending forward.
  Arms: Diaphragm hipopressive exercise
Other: Ischemic compression techniques in shoulder myofascial trigger points — Ischemic compression techniques in infraespinatus and supraespinatus myofascial trigger points during one minute each muscle. The pressure increases gradually until the individual feels a tolerable pain.
  Arms: Shoulder myofascial trigger points treatment

SUMMARY:
A randomised and controlled trial to people diagnosed with rotator cuff injuries who are divided into 3 groups of treatment: shoulder myofascial trigger points release, manual diaphragm release and diaphragm mobilization through hipopressive gymnastic exercise. The pain and range of shoulder movement are assessed before and after the treatment in all the participants.

Hypothesis of the clinical study: the treatment of diaphragm muscle, via manual release or active mobilization, has impact on rotator cuff injury symptoms comparing with a standard treatment of shoulder myofascial trigger points release.

Discussion: The relation between shoulder and diaphragm muscle, through innervation (phrenic nerve and brachial plexus), embryology and myofascial connections, could lead to include in clinical practice the examination and treatment of other structures besides shoulder girdle such as diaphragmatic region in rotator cuff injuries.

DETAILED DESCRIPTION:
This study is a randomised controlled trial evaluating clinical effects of a diaphragm treatment, via manual release or active mobilization, comparing with a standard treatment of shoulder myofascial trigger points release.

A description of the 3 groups of treatment:

1. - Experimental group 1: 3 diaphragm stretching techniques according to Chaitow, Ward and Ricard, performed by a physical therapist are employed in this experimental group during 10 minutes. The participants are situated in a seated, supine and side bending position.
2. - Experimental group 2: diaphragm mobilization through active hipopressive gymnastic exercise according to Caufriez in two different postures.
3. - Active comparator group: A ischemic compression technique in most painful myofascial trigger points in the infraespinatus and supraespinatus muscle during one minute each one.

The shoulder flexion, abduction and external rotation range of motion will be assessed pre and postinterventions, as well as the pressure pain threshold with an algometer and the pain experienced by the individual in shoulder mobility with a Numerical Rating Scale.

ELIGIBILITY:
Inclusion Criteria:

* Participants of both genders aged between 18 and 65 years old
* Ultrasound and/or magnetic resonance imaging diagnosis of rotator cuff injury
* Pain or range of movement restriction in active shoulder flexion and/or abduction

Exclusion Criteria:

* Use of analgesic or anti-inflammatory drugs 72 hours prior to the study
* Individuals with glenohumeral instability due to shoulder luxation or subluxation or Bankart labrum injury
* Individuals who have received physical therapy treatment in last week
* Individuals who underwent thoracic or shoulder surgery or people suffering from rheumatisms
* Diabetic patients
* People with a diagnosed neurological pathology
* Individuals with a diagnosed mental health problem
* Not being able to understand and sign the informed consent and information sheet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline to post intervention shoulder range of motion with a digital inclinometer | Baseline and Immediately Post Intervention
  Pre and post treatment assessment of flexion, abduction and external rotation at 90º abduction movements in supine, registered with a Baseline digital inclinometer
Change from baseline to post intervention pressure pain threshold in supraespinatus tendon and xiphoid process with a pressure algometer | Baseline and Immediately Post Intervention
  Pre and post treatment Pressure pain threshold in supraespinatus tendon and xiphoid process registered with a pressure algometer in a supine position
Change from baseline to post intervention Numerical Rating Pain Scale in shoulder mobility | Baseline and Immediately Post Intervention
  Pre and post treatment Numerical Rating Pain Scale in shoulder mobility: flexion, abduction and external rotation at 90º abduction standing

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Complutense de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2017-11-24): https://cdn.clinicaltrials.gov/large-docs/29/NCT03293329/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-24): https://cdn.clinicaltrials.gov/large-docs/29/NCT03293329/SAP_001.pdf